CLINICAL TRIAL: NCT04847284
Title: Intraoperative Radiotherapy in Patients With Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/9548/I
Record Dates: First submitted 2021-03-25; First posted 2021-04-19 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-10

CONDITIONS: Brain Metastases
Keywords: Brain metastases; Intraoperative radiotherapy; Intrabeam
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arms (Experimental): To determine the efficiency and safety of IORT with low-energy photons to the cavity after resection of brain metastases
  Interventions: Radiation: Intraoperative radiotherapy

INTERVENTIONS:
Radiation: Intraoperative radiotherapy — Intraoperative radiotherapy application immediately following resection of brain metastases.

SUMMARY:
Intraoperative radiotherapy (IORT) is a new alternative for local radiotherapy with the advantages of dose escalation, reduced overall treatment time, and enhanced patient convenience, however the degree of efficacy is unknown, as well as and which is the most efficient dose.

The objective of this study is to evaluate the efficacy and safety of IORT in patients with surgical excision of brain metastases at a dose of 20 Gy is at least as effective and safe as other forms of radiation therapy in patients with resection of brain metastases.

DETAILED DESCRIPTION:
1. INTRODUCTION

   Brain metastases occur in roughly 30% of all cancer patients during their course of disease. Their incidence is believed to rise due to the aging population that develops more cancer per se, an increase in overall survival due to more effective extracranial therapies but with only few (novel) substances crossing the blood-brain barrier and more broadly available and more advanced imaging techniques.

   Neurosurgical treatment remains a cornerstone in the management of brain metastasis, especially for lesions causing mass effects or neurological deficits or in case tissue is necessary to establish a diagnosis. As local recurrence rates are as high as 50-60% after surgical resection alone, adjuvant therapies to prevent such are necessary.

   Whole brain radiotherapy (WBRT) does not influence survival but rather impairs neurocognitive functions and, as histologic in-depth exams of cavity borders showed that most brain metastases infiltrate only 0.3-1.2 mm into the surrounding healthy brain tissue, therefore treatment is to date usually confined to the cavity margin. Thus, the currently recommended standard of care is post-operative stereotactic radiosurgery (SRS) to the resection cavity. One of the drawbacks of this modality is the incidence of radionecrosis, especially in large tumor volumes. As an alternative to radiosurgery, hypofractionated local radiotherapy is also used, reducing the risk of radionecrosis in large volumes. There are no prospective randomized studies comparing both techniques.

   The need to find a modality of radiotherapy that achieves al least the efficacy of radiosurgery or hypofractionated local radiotherapy, without the disadvantages thereof, makes IORT as a possible treatment alternative.

   The objective of this study is to evaluate the efficacy and safety of IORT in patients with surgical excision of brain metastases at a dose of 20 Gy is at least as effective and safe as other forms of radiation therapy in patients with resection of brain metastases.
2. OBJECTIVES

   Primary Objective
   * Median local progression free survival (lPFS), defined as time span (in months) between surgery and recurrence within a 0,5 cm margin around the resection cavity, assessed by serial MRI scans and RANO response assessment criteria for brain metastases .
   * Radiation-related (acute / late) neurotoxicity, assessed by regular neurological examinations and serial MRI scans.

   Secondary objectives
   * Median regional PFS (rPFS), resembling the time (in months) from surgery to any progression outside of the 0,5 cm margin around the resection cavity, assessed by serial MRI scans and RANO response assessment criteria for brain metastases .
   * Global PFS (gPFS), defined as the time (in months) from surgery to any intra- and extracranial tumor progress.
   * Median overall survival (OS), defined as the time (in months) from surgery of brain metastases to death from by any cause.
3. DESIGN

This trial is an open, single arm, single institution, prospective trial to determine the efficiency and safety of IORT with low-energy photons to the cavity after resection of brain metastases. A total of 25 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Karnofsky Performance Status ≥ 70
* Newly diagnosed cerebral or cerebellar lesion (contrast enhancing on a T1-weighted MRI scan) amenable to total resection with no dural attachment
* Frozen section confirming a metastasis of an extracranial ( Central Nervous System i.e. non-CNS) tumor
* Adequate distance to optic nerve(s), chiasm and brainstem (organs at risk for radiotherapy)
* Adequate birth control

Exclusion Criteria:

* Leptomeningeal spread and dural attachment (assessed pre- and intraoperatively)
* Frozen section reveals primary CNS tumor, lymphoma, SCLC (Small-cell lung cancer) or germinoma
* More than one brain metastasis
* Psychiatric or social condition potentially interfering with compliance
* Contraindication against anesthesia, surgery, MRI and/or contrast agents
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Median local progression free survival (lPFS) | 6 months from the date of surgery.
  Recurrence within a 0.5 cm margin around the resection cavity, assessed by serial magnetic resonance imaging (MRI scans) and response assessment criteria in neuro-oncology (RANO)
Radiation-related acute neurotoxicity | 3 months from the date of surgery.
  Neurotoxicity related to radiotherapy evaluated according to the scale of the Common Terminology Criteria for Adverse Events (CTCAE) version 5. Score from 0 to 5, with 5 being the worst toxicity
  - Acute toxicity: cerebral edema
Radiation-related late neurotoxicity | 6 months from the date of surgery.
  Neurotoxicity related to radiotherapy evaluated according to the scale of the Common Terminology Criteria for Adverse Events (CTCAE) version 5. Score from 0 to 5, with 5 being the worst toxicity
  - Late toxicity: radionecrosis.

SECONDARY OUTCOMES:
Median regional PFS (rPFS) | 6 months from the date of surgery
  To any progression outside of the 0.5 cm margin around the resection cavity, assessed by serial MRI scans and RANO response assessment in neuro-oncology .
Global PFS (gPFS) | 6 months from the date of surgery
  The time (in months) from surgery to any intra- and extracranial tumor progress
Median overall survival (OS) | 6 months from the date of surgery
  The time (in months) from surgery of brain metastases to death from by any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giordano FA, Brehmer S, Murle B, Welzel G, Sperk E, Keller A, Abo-Madyan Y, Scherzinger E, Clausen S, Schneider F, Herskind C, Glas M, Seiz-Rosenhagen M, Groden C, Hanggi D, Schmiedek P, Emami B, Souhami L, Petrecca K, Wenz F. Intraoperative Radiotherapy in Newly Diagnosed Glioblastoma (INTRAGO): An Open-Label, Dose-Escalation Phase I/II Trial. Neurosurgery. 2019 Jan 1;84(1):41-49. doi: 10.1093/neuros/nyy018. PMID 29528443
- [Result] Weil RJ, Mavinkurve GG, Chao ST, Vogelbaum MA, Suh JH, Kolar M, Toms SA. Intraoperative radiotherapy to treat newly diagnosed solitary brain metastasis: initial experience and long-term outcomes. J Neurosurg. 2015 Apr;122(4):825-32. doi: 10.3171/2014.11.JNS1449. Epub 2015 Jan 23. PMID 25614945
- [Result] Cifarelli CP, Brehmer S, Vargo JA, Hack JD, Kahl KH, Sarria-Vargas G, Giordano FA. Intraoperative radiotherapy (IORT) for surgically resected brain metastases: outcome analysis of an international cooperative study. J Neurooncol. 2019 Nov;145(2):391-397. doi: 10.1007/s11060-019-03309-6. Epub 2019 Oct 25. PMID 31654248
- [Result] Vargo JA, Sparks KM, Singh R, Jacobson GM, Hack JD, Cifarelli CP. Feasibility of dose escalation using intraoperative radiotherapy following resection of large brain metastases compared to post-operative stereotactic radiosurgery. J Neurooncol. 2018 Nov;140(2):413-420. doi: 10.1007/s11060-018-2968-4. Epub 2018 Aug 9. PMID 30094718